CLINICAL TRIAL: NCT03232086
Title: Responses to Exposure to Low Levels of Concentrated Ambient Particles in Healthy Young Adults
Acronym: RECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Diaz-Sanchez, Chief, Clinical Research Branch, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-1548
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Exposure to Pollution
Keywords: Controlled Human Exposure Study; Cardiovascular
MeSH Terms: interventions — Environment, Controlled

STUDY DESIGN:
Intervention Model Description: Clean Air
  Concentrated PM2.5
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clean Air (Sham Comparator): Exposure to clean air will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus.
  Interventions: Other: Clean Air
- Concentrated PM2.5 (Active Comparator): Exposure to PM2.5 will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus.
  Interventions: Other: PM2.5

INTERVENTIONS:
Other: Clean Air — Each subject will be exposed to clean air for 4 hours. Subjects will exercise on a bike or treadmill. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/min/m2BSA followed by a 15 minute rest period.
  Arms: Clean Air
Other: PM2.5 — Each subject will be exposed up to 35-50 μg/m3 PM2.5 for 4 hours. Subjects will exercise on a bike or treadmill. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/min/m2BSA followed by a 15 minute rest period.
  Arms: Concentrated PM2.5

SUMMARY:
Purpose: To determine whether exposure to levels of fine particles that are close to the current standard will cause cardiovascular changes in healthy individuals.

DETAILED DESCRIPTION:
Air pollution is associated with several adverse health outcomes. Specifically, ambient fine particulate matter ≤2.5 μg/m3 (PM2.5) is associated with increased mortality and increased risk for respiratory and cardiovascular disease It has been estimated that worldwide over 3.2 million premature deaths and over 74 million years of healthy life lost were attributable to ambient particulate matter pollution, making it one of the top global health risk factors . Further, an estimated 22% of disability-adjusted life-years for heart disease are attributable to ambient particulate matter pollution. Similarly, it is estimated that air pollution exposure contributed to about 6% (3.7 million) of all deaths in 2012, with 40% of those coming from coronary artery disease (CAD). More than 100 time-series and case-crossover analyses have demonstrated associations of short term PM2.5 exposure with myocardial infarctions (MIs); aggravated asthma and increased risk for hospitalizations and mortality. These studies suggest that the acute health effects of air pollution particularly affect infants and children, older adults, and those with underlying disease, such as diabetes and cardiovascular disease (Pope, 2014). In healthy and younger individuals (<65 year old) these same studies observe associations between air pollution and subclinical biomarkers of inflammation, coagulation and oxidative stress but not for any clinical outcomes. This has led the American Heart Association to state that" Despite theoretical statistical risks ascribed to all individuals, this elevated risk from exposure is not equally distributed within a population. At present-day levels, PM2.5 likely poses an acute threat principally to susceptible people, even if seemingly healthy, such as the elderly and those with (unrecognized) existing coronary artery or structural heart disease."

Controlled human exposure studies are a critical component of the health risk assessment for ozone because of their ability to establish exposure-response relationships at low doses and have therefore weighed heavily in deliberations when the U.S. EPA has considered the National Ambient Air Quality Standard (NAAQS). In contrast, for PM2.5, controlled exposure studies have been used primarily to demonstrate biological plausibility. that is the potential for particulate matter to exert extra-pulmonary effects. These studies have shown that healthy volunteers primarily exhibit mild pulmonary inflammation, decreases in heart rate variability and changes in blood factors associated with blood coagulation following exposure to concentrated air particles (CAPs), most show no change in lung function and none result in cardiac arrhythmia. Nearly all these studies have been conducted at realistic but high levels of PM2.5 (typically above 100 µg/m3). Currently the EPA 24-hour fine particle standard is 35µg/m3, a value based predominantly on epidemiologic studies. While epidemiologic studies suggest that similar effects can occur at lower levels, it is difficult for these association studies to conclusively demonstrate because of the problems in disassociating the effects of PM2.5 from other pollutants and confounders. Only a controlled human exposure study can determine directly whether PM2.5 can alter cardiovascular endpoints at lower concentrations. Four hours represents a typical exposure duration to particulate matter during the course of the day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals ages 18-35 years of age
* Physical conditioning allowing intermittent, moderate exercise for four hours. Ability to complete the exposure exercise regimen without reaching 80% of predicted maximal heart rate. Predicted maximal heart rate will be calculated using the equation (described by Tanaka et al.: [2001] J. Am. Coll. Cardiol.): [208bpm-((0.7) x (age in years))]
* Normal baseline 12-lead EKG .
* Normal lung function

  1. Forced vital capacity (FVC) ≥ 80% of that predicted for gender, ethnicity, age and height (according to NHANESIII guidelines).
  2. Forced expiratory volume in one second (FEV1) ≥ 80%of that predicted for gender,ethnicity, age and height
  3. FEV1) /FVC ratio≥ 80% of predicted values.
* Oxygen saturation ≥ 96% on room air.

Exclusion Criteria:

* Individuals with a history of acute or chronic cardiovascular disease, chronic respiratory disease, diabetes, rheumatologic diseases, or immunodeficiency state.
* Individuals with a CVD risk score greater than 10% using the ACC/AHA ASCVD risk calculator.
* Individuals with clinically diagnosed asthma.
* Individuals who are allergic to chemical vapors or gases.
* Females who are pregnant, attempting to become pregnant, or breastfeeding.
* Individuals that are unable or unwilling to stop for at least two weeks prior to the study taking medications, vitamins or supplements that the investigators believe may impact the results of the study. Those not specifically mentioned here may be reviewed by the investigators prior to an individual's inclusion in the study.
* Individuals who smoke/vape more than 2 times per month and have smoked/vaped within 4 weeks prior to all study visits.
* Individuals living with a smoker who smokes inside the house.
* Individuals with a body mass index (BMI) >35 or <18. Body mass index is calculated by dividing the weight in kilograms by the square of the height in meters.
* Individuals with occupational exposures to high levels of vapors, dust, gases, or fumes on an on-going basis.
* Individuals with uncontrolled hypertension (≥150 systolic or ≥90 diastolic).
* Individuals that do not understand or speak English.
* Individuals that are unable to perform the exercise required for the study.
* Individuals that are taking beta blocker medications.
* Individuals with a history of skin allergies to adhesives used in securing EKG electrodes.
* Individuals with unspecified diseases, conditions, or medications that might influence the responses to the exposures, as judged by the medical staff.
* Individuals that are unwilling or unable to stop taking over-the-counter pain medications such as aspirin, ibuprofen (Advil, Motrin), naproxen (Aleve), or other non-steroidal anti-inflammatory ("NSAID") medications for 48 hours prior to the exposures and post-exposure visits.
* Individuals that are taking systemic steroids or beta-blocker medications.
* Individuals with a hemoglobin A1c (HbA1c) level > 6.4%.

Temporary Exclusion Criteria:

* Individuals suffering from acute respiratory illness within four weeks prior to any of the study exposure series.
* Individuals that have been exposed to smoke and fumes within 24 hours of any study visit.
* Individuals that have engaged in strenuous exercise within 24 hours of any study visit.
* Individuals that have been exposed to ozone-based home air purifiers within 24 hours of any study visit.
* Individuals unable to avoid drinking alcohol for 24 hours prior to all study visits.
* Individual unable to avoid caffeine for 12 hours prior to all study visits and during each study visit.
* Individuals that have been exposed to unvented household combustion sources (gas stoves, lit fireplaces, oil/kerosene heaters) within 48 hours of any study visit.
* Individuals that have been exposed to or have consumed any agent or have undertaken any activity within 24 hours of any study visit that the investigators believe may compromise the results of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate variability | Pre exposure to 24hours post exposure
  10 minute electrocardiogram recording (measured by Holter ECG) in which the

SECONDARY OUTCOMES:
Forced expired volume in the first second (FEV1) | Pre exposure to 24hours post exposure
  Forced expired volume in the first second (FEV1) is determined by spirometry performed on a dry seal spirometer interfaced to a computer.
Forced Vital Capacity | Pre exposure to 24hours post exposure
  Forced Vital Capacity(FVC) is determined by spirometry performed on a dry seal spirometer interfaced to a computer.
Index of inflammatory markers | Pre exposure to 24hours post exposure
  Index of inflammatory markers is the mean % changes in a basket of factors related to systemic inflammation (IL-6, IL-8, TNF-a, IL-b, CRP) in the blood following exposure to PM2.5 vs. clean air.

CONTACTS AND LOCATIONS:
Locations (1):
- U.S. EPA Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Derived] Wyatt LH, Devlin RB, Rappold AG, Case MW, Diaz-Sanchez D. Low levels of fine particulate matter increase vascular damage and reduce pulmonary function in young healthy adults. Part Fibre Toxicol. 2020 Nov 16;17(1):58. doi: 10.1186/s12989-020-00389-5. PMID 33198760